CLINICAL TRIAL: NCT04464343
Title: The Biomechanical Mechanism for Gait and Plantar Pressure Changes After Posterior Cruciate Ligament Rupture and Reconstruction
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OR006
Record Dates: First submitted 2020-06-29; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Posterior Cruciate Ligament Tear
Keywords: posterior cruciate ligament; knee; hip; ankle; biomechanics; walking; jogging; cutting; jumping

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Posterior cruciate ligament injury group: According to the previous clinical diagnosis, volunteers who has never suffered the Posterior cruciate ligament injury.
  Interventions: Other: no intervention
- normal control group: According to the previous clinical diagnosis, volunteers who has never suffered the lower extremity sports injuries.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This is an observation study, with no intervention

SUMMARY:
Investigating the biomechanics for the PCL ruptured or reconstructed patients during walking, jogging, cutting, jumping. To establish a knee joint biomechanical evaluation model to quantify and evaluate the plantar pressure information under dynamic load-bearing state after PCL fracture. Provide a precise basis for the biomechanical state of the knee, and establish a clinically practical automatic analysis of plantar pressure information and an expert diagnostic system.

DETAILED DESCRIPTION:
Background: The posterior cruciate ligament (PCL) is an essential structure in knee stabilization. Knee cartilage degeneration after a PCL injury has been reported in several studies. Understanding the changes in movement patterns of patients with PCL ruptures could help clinicians make specific treatment protocols to restore patients' sporting ability and prevent joint degeneration. However, the kinematics and kinetics of the lower limb in patients with PCL injuries are still not clear.

Methods: Three-dimensional gait analysis system, force plate, electromyography will be used for 55 healthy male participants (control group) and 55 male patients with isolated PCL-deficiency (PCL-d group) during walking, jogging, cutting, jumping. Repeated measurement two-factor analysis of variance will be performed to determine differences between involved and uninvolved legs in the PCL-d group and control group at different rehabilitation times (prior reconstruction surgery, 6 months, and 1-year post PCL reconstruction surgery). Three-dimensional gait analysis and computer-aided analysis technology of plantar pressure information were used to study the changes of PCL after fracture and reconstruction. Based on the plantar pressure information, the movement parameters, and individual attribute parameters, establish a knee joint biomechanical evaluation model to quantify and evaluate the plantar pressure information under dynamic load-bearing state after PCL fracture. Provide a precise basis for the biomechanical state of the knee, and establish a clinically practical automatic analysis of plantar pressure information and an expert diagnostic system.

ELIGIBILITY:
Inclusion Criteria:

* age of 18-45 years old
* Isolated PCL rupture patients: The inclusion criteria included an isolated PCL rupture of at least 3 months' duration.
* Healthy volunteers: no history of neuro or musculoskeletal system injury that may affect the movements.

Exclusion Criteria:

* additional knee ligament or meniscal damage
* severe damage to the ipsilateral hip, ankle joint, or contralateral lower limb (ligament ruptures or bone fractures)
* age >50 years (to avoid age-induced osteoarthritis interference)
* any cartilage injury grade >2 according to the Outerbridge classification
* Tegner score18 <3

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Inclusion：age of 18-45 years old. Healthy volunteers: no history of neuro or musculoskeletal system injury that may affect the movements. Isolated PCL rupture patients: The inclusion criteria included an isolated PCL rupture of at least 3 months' duration. The exclusion criteria were (1) additional knee ligament or meniscal damage; (2) severe damage to the ipsilateral hip, ankle joint, or contralateral lower limb (ligament ruptures or bone fractures); (3) age >50 years (to avoid age-induced osteoarthritis interference); (4) any cartilage injury grade >2 according to the Outerbridge classification; and (5) Tegner score18 <3.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2014-06-14 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
walking speed | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
ground reaction force | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
knee flexion angle | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
the moment of knee extension in the gait cycle | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.
the moment of knee flexion in the gait cycle | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking, jogging, cutting and jumping.

SECONDARY OUTCOMES:
The International Knee Documentation Committee (IKDC) score | On the day of enrollment.
  The International Knee Documentation Committee (IKDC) score was used to evaluate the knee health.The patients completed score by themselves. The lowest score is 0 and the highest score is 100. The higher is better.

CONTACTS AND LOCATIONS:
Overall Officials: Hongshi Huang, Doctor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No